CLINICAL TRIAL: NCT06170008
Title: Efficacy of a Transparent Silicone Membrane With Physical Microstructure for Second-degree Burn Wounds and Skin Graft Wounds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: chhaodylan
Record Dates: First submitted 2023-06-04; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Second-degree Burn Wounds; Skin Graft Wounds
Keywords: Second-degree burn wounds; skin graft wounds; Wound coverings

STUDY DESIGN:
Intervention Model Description: The second-degree burn wounds were covered with clear silicone film and decellularized pig skin after conventional clinical treatment.
  After skin grafting, the wounds were covered with transparent silicone film and petroleum jelly gauze with physical microstructure modification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Second-degree burn wounds covered with silicone film sheet group (Experimental): After routine clinical treatment of second-degree burn wounds, the innermost layer is covered with physical microstructure-modified transparent silicone film sheet , and the outer dressing is changed every 3 to 4 days to observe and record the wounds, and the innermost dressing is changed weekly or as necessary and the number of times is recorded to observe the wound healing rate, dressing transparency, dressing-wound adhesion, pain level, wound infection rate and incidence of adverse reactions.
  Interventions: Device: Physical microstructure-modified transparent silicone film sheet
- Second-degree burn wounds covered with decellularized pig skin group (Active Comparator): After routine clinical treatment of second-degree burn wounds, the innermost layer was covered with decellularized pig skin, the outer dressing was changed every 3 to 4 days, the wounds were observed and recorded, and the innermost dressing was changed weekly or as necessary and the number of times was recorded to observe the wound healing rate, dressing transparency, dressing-wound adhesion, pain level, wound infection rate and incidence of adverse reactions.
  Interventions: Device: Decellularized pig skin
- Post-operative skin grafting wounds covered with silicone film sheet group (Experimental): After skin grafting, the innermost layer is covered with physical microstructure-modified transparent silicone film sheet , and the outer dressing is changed every 3 to 4 days to observe and record the wound. The innermost layer is changed weekly or as necessary and the number of times is recorded to observe the wound healing rate, transparency of the dressing, adhesion of the dressing to the wound, pain, wound infection rate and incidence of adverse reactions.
  Interventions: Device: Physical microstructure-modified transparent silicone film sheet
- Post-operative skin grafting wounds covered with vaseline gauze group (Active Comparator): After skin grafting, the innermost layer was covered with vaseline gauze, and the outer layer was changed every 3 to 4 days to observe and record the wound. The innermost layer was changed weekly or as necessary and the number of times was recorded to observe the wound healing rate, transparency of the dressing, adhesion of the dressing to the wound, pain, wound infection rate and incidence of adverse reactions.
  Interventions: Device: Vaseline gauze

INTERVENTIONS:
Device: Physical microstructure-modified transparent silicone film sheet — The main component of the physical microstructure-modified transparent silicone film sheet is transparent silicone rubber, which has a three-dimensional microstructure on its trauma contact surface through physical mechanics treatment, which can provide effective mechanical stimulation for trauma healing. And after testing, the silicone film sheet is breathable, light-permeable, non-toxic and non-allergenic. It is expected to significantly reduce the number of dressing changes, reduce the damage to the wound and the painful stimulation to the patient during dressing changes, and promote the healing of the wound to a certain extent, thus improving the quality of wound repair and saving medical costs.
  Arms: Post-operative skin grafting wounds covered with silicone film sheet group; Second-degree burn wounds covered with silicone film sheet group
Device: Decellularized pig skin — Decellularized pig skin is an allogeneic trauma covering from pigs and is a commonly used trauma covering for second-degree burn wounds. It adheres to clean superficial wounds, creates a temporary barrier to the wound, reduces wound exudation, limits loss of body components, improves microcirculatory stasis, provides a microenvironment suitable for wound healing, protects inter-ecological tissue, promotes repair and regeneration, and reduces pain. Its disadvantages are: soft structure, difficult to fix the trauma; opaque, unable to observe the trauma; pigskin needs to be stored under suitable temperature and humidity, and has a limited time. When used, decellularized pig skin is directly covered on conventionally treated second-degree burn wounds.
  Arms: Second-degree burn wounds covered with decellularized pig skin group
Device: Vaseline gauze — Vaseline gauze is the most commonly used conventional dressing for the implant area, which is mainly made of skimmed cotton gauze impregnated with petroleum jelly and paraffin oil, which has a lubricating effect and can promote the growth of granulation and wound healing. However, its moisturizing time is relatively short and requires frequent dressing changes; moreover, petroleum jelly gauze often adheres to the wound surface severely, which may cause bleeding and new epidermal damage during dressing changes and affect the wound healing; the wound surface is constantly oozing blood and fluid, and the dressing cannot be effectively isolated from the outside world after wetting, which increases the chance of infection. Vaseline gauze is applied directly to the post-operative skin grafting wound.
  Arms: Post-operative skin grafting wounds covered with vaseline gauze group

SUMMARY:
The goal of this clinical trial is to comparison of physical microstructure-modified transparent silicone films and current conventional trauma dressings for second-degree burn wounds and post-skin graft wounds.The main question it aims to answer is :

The development of a new type of wound dressing is urgently needed because existing wound dressings cannot be transparent, easy to change, easy to store and inexpensive at the same time.

Participants will receive routine wound treatment, after which they will be covered with a clear silicone membrane with physical microstructure modification.

Researchers will compare vaseline gauze group and decellularised pigskin group o see if transparent silicone film with physical microstructure modifications promotes wound healing, reduces the number of dressing changes, reduces the damage to the wound and painful irritation to the patient during dressing changes, thus improving the quality of wound repair and saving medical costs.

DETAILED DESCRIPTION:
In this study, a single-centre, autologous petrolatum gauze or decellularised pig skin treatment was used to study the effect of physical microstructure-modified transparent silicone membranes on the repair of second-degree burn wounds and implant-area wounds in a parallel controlled study using a randomised controlled clinical trial. In this study, 40 patients were enrolled in the burn surgery department of the First Affiliated Hospital of the Naval Military Medical University, with 20 second-degree burn wounds and 20 implant-area wounds each. The same patients were divided into a conventional treatment group (second-degree burn wounds covered with decellularized pig skin and implant-area wounds covered with petroleum jelly gauze) and a silicone film-covered group according to the computerized random number method. After routine clinical treatment of the wounds, the wounds were covered with the corresponding dressings according to the groups, and the healing rate, transparency of the dressings, adhesion of the dressings to the wounds, pain level of the patients when the dressings were removed, infection rate of the wounds and incidence of adverse reactions were observed.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 70 years, regardless of gender;
* Second-degree burns with an area greater than 1% TBSA and a single observable trauma area ≥ 10 cm × 10 cm(jointly determined by two burn specialists with the title of attending physician or above according to the four degrees and five points method);
* Voluntary signed informed consent form

Exclusion Criteria:

* Patients during pregnancy;
* Significant cardiac, pulmonary and renal insufficiency;
* Critically ill or with serious complications such as severe sepsis or MODS;
* Positive for HBV, HCV, HIV or syphilis;
* Traumatic surface infection;
* Involving the face, hands, groin, joints, feet and other areas difficult to bandage and fix; previous burn trauma treatment; previous burns on the same site; electrical burns; patients with inhalation injuries.
* Known sensitivity or allergy to one of the dressings or its components; diabetes mellitus; presence of immune system disorders or long-term hormone or immunotherapy
* Others who, in the opinion of the investigator, are not suitable for enrollment.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing time | one day interval after wound coverage application
  Change the dressing at one-day intervals after the application of trauma coverings, observe the trauma, and record the healing time when the trauma is 90% healed. The wound healing rate is: healed wound area / original wound area. There are two methods to calculate the healed area: A, visual method: visual assessment; B, image analysis method: vertical trauma surface is photographed under natural light (20CM and 40CM respectively), and the computer analyzes the trauma healing rate. The image analysis method shall prevail, and the image method shall prevail in case of inconsistent results.
Wound healing rate | 14th days after the treatment
  The wound healing rate was calculated on the 14th days after the treatment. The wound healing rate was calculated as: healed wound area/ original wound area. There are two methods for calculating the healed area: A, visual method: visual assessment; B, image analysis method: vertical trauma surface is photographed under natural light (20CM and 40CM distance respectively) and the computer analyzes the trauma healing rate. The image analysis method shall prevail, and the image method shall prevail in case of inconsistent results.

SECONDARY OUTCOMES:
Transparency | 7th, 14th, 21st and 28th days after the treatment
  The transparency of the inner dressing was evaluated at days 7, 14 after wound treatment. They were: clear, the trabecular base could be observed (including fluid infection, survival of trabecular new epithelium or graft, etc.); obscure, the trabecular base was faintly visible; opaque, the trabecular base could not be observed.
Adhesions and pain | 7th, 14th, 21st and 28th days after the treatment
  Observe the degree of adhesion and patient pain when changing the inner dressing. Scoring using the "Changhai Pain Ruler", with 0 indicating no pain; 1~3 indicating slight pain, tolerable; 4~6 indicating obvious pain and affecting sleep, still tolerable; 7~10 indicating strong pain, affecting appetite for sleep, unbearable.
Number of inner layer dressing changes | Within four weeks of treatment
  Record the number of inner dressing changes during the wound healing process.
Infection rate | 7th, 14th, 21st and 28th days after the treatment
  Wound infection was observed at 7, 14, 21, and 28 days after transplantation, respectively.Observation of trauma infection: amount and nature of trauma secretion, odor; peri-trauma skin temperature and presence of redness, swelling and pressure pain.
  Bacterial culture of trauma secretions: Bacterial culture of secretions was performed at 7, 14 and 21 days after transplantation.
Incidence of adverse reactions | 7th, 14th, 21st and 28th days after the treatment
  Observe for the development of variant contact dermatitis (ACD), i.e., extensive pruritus, eczema-like lesions, and positive patch test.